CLINICAL TRIAL: NCT00003238
Title: A Phase II Trial of Perillyl Alcohol (NSC 641066) Administered Daily In Patients With Metastatic Androgen Independent Prostate Cancer
Brief Title: Perillyl Alcohol in Treating Patients With Metastatic Prostate Cancer That Has Not Responded to Hormone Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000066113; R03CA073906 (NIH); WCCC-CO-9685; NCI-T97-0067
Record Dates: First submitted 1999-11-01; First posted 2004-07-21 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2013-08

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — perillyl alcohol

INTERVENTIONS:
Drug: perillyl alcohol

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different way to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of perillyl alcohol in treating patients with metastatic prostate cancer that has not responded to hormone therapy with androgens.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the clinical effectiveness of oral perillyl alcohol given to patients with androgen independent metastatic prostate cancer. II. Assess the toxicity of this treatment in these patients.

OUTLINE: Patients receive oral perillyl alcohol 4 times a day for 4 weeks. Patients continue treatment in the absence of severe toxicity and disease progression. Patients are followed every 3 months for survival after disease progression.

PROJECTED ACCRUAL: This study will accrue 20-40 patients in approximately 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed progressive metastatic or progressive regional nodal adenocarcinoma of the prostate Regression of tumor following hormone therapy If on antiandrogen therapy, must fail to respond to withdrawal or have progressive disease following withdrawal of antiandrogen No CNS disease

PATIENT CHARACTERISTICS: Age: Not specified Performance status: WCCC 0-2 Life expectancy: At least 3 months Hematopoietic: WBC at least 3000/mm3 Absolute neutrophil count at least 1200/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 8 g/dL Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT no greater than 2.5 times normal Renal: Creatinine no greater than 1.5 times upper limit of normal Other: At least 5 years since prior malignancy other than: Inactive nonmelanoma skin cancer Adequately treated stage I or II cancer in complete remission No other serious illness No spinal cord compression symptoms

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Prior chemotherapy required Endocrine therapy: Failed one secondary hormonal manipulation for metastatic disease Concurrent testicular androgen suppression (LHRH) allowed No concurrent hormonal therapy other than LHRH agonist At least 4 weeks since antiandrogen treatment in order to evaluate for response withdrawal Radiotherapy: At least 4 weeks since prior radiation therapy No prior strontium therapy Surgery: No prior orchiectomy Other: No concurrent cholesterol lowering agents No concurrent supplemental vitamins No concurrent antioxidants

Max Age: 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-02; Primary Completion 2001-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Wilding, MD, Study Chair — University of Wisconsin, Madison
Locations (8):
- United States (8):
  - Leonard C. Ferguson Cancer Center, Freeport, Illinois
  - Green Bay Oncology, Ltd., Green Bay, Wisconsin
  - Mercy Health System, Janesville, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Meriter Hospital, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Sinai Samaritan Medical Center - Milwaukee, Milwaukee, Wisconsin
  - North Central Oncology Associates, S.C., Wausau, Wisconsin